CLINICAL TRIAL: NCT02680561
Title: A Double-Blind (Incorporating an Open Label Comparator), 3-Period, Crossover Study to Determine the Pharmacokinetic Profile and Tolerability of Single Doses of Fluticasone Propionate Multidose Dry Powder Inhaler and Fluticasone Propionate/Salmeterol Multidose Dry Powder Inhaler Compared to ADVAIR® DISKUS® in Patients With Persistent Asthma 4 Through 11 Years of Age
Brief Title: A Double Blind Open Label Comparator Study to Compare Treatments in 4 to 11 Year Old Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FSS-PK-10007
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: Fp MDPI (Experimental): Single inhalation dose of Fluticasone Propionate Multidose Dry Powder Inhaler (Fp MDPI) on Day 1 into 1 of 6 treatment sequences (ABC, BCA, CAB, ACB, BAC, or CBA)
  Interventions: Drug: Fluticasone Propionate MDPI; Drug: Fluticasone Propionate/Salmeterol MDPI; Drug: Fluticasone propionate/salmeterol
- Treatment B: FS MDPI (Experimental): Single inhalation dose of Fluticasone Propionate/Salmeterol Multidose Dry Powder Inhaler (FS MDPI) on Day 1 into 1 of 6 treatment sequences (ABC, BCA, CAB, ACB, BAC, or CBA)
  Interventions: Drug: Fluticasone Propionate MDPI; Drug: Fluticasone Propionate/Salmeterol MDPI; Drug: Fluticasone propionate/salmeterol
- Treatment C: Comparator (Active Comparator): Single inhalation dose of fluticasone propionate/salmeterol (ADVAIR DISKUS) on Day 1 into 1 of 6 treatment sequences (ABC, BCA, CAB, ACB, BAC, or CBA)
  Interventions: Drug: Fluticasone Propionate MDPI; Drug: Fluticasone Propionate/Salmeterol MDPI; Drug: Fluticasone propionate/salmeterol

INTERVENTIONS:
Drug: Fluticasone Propionate MDPI
  Other Names: Fp MDPI
Drug: Fluticasone Propionate/Salmeterol MDPI
  Other Names: FS MDPI
Drug: Fluticasone propionate/salmeterol
  Other Names: ADVAIR; DISKUS

SUMMARY:
The purpose of the study is to characterize the pharmacokinetic profiles of fluticasone propionate and/or salmeterol when delivered as a single oral inhalation dose of Fp MDPI and FS MDPI.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male or female aged 4 through 11 years of age, inclusive
* Severity of disease: The patient has persistent asthma
* Asthma diagnosis: The patient has a diagnosis of asthma as defined by the NIH.
* The patient has required less than 4 inhalations per week of rescue bronchodilator (on average) for the 4 weeks preceding the SV.
* The patient is able to withhold (as judged by the investigator) his or her rescue medication for at least 6 hours before the SV and before all treatment visits.
* The patient must have a weight of 18 kg or higher.

  * Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* The patient has a history of a life-threatening asthma exacerbation that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, or hypoxic seizures.
* Female patients that have reached puberty and have a child bearing potential must have a negative serum pregnancy test at the SV. Eligible menstruating female patients unwilling to employ appropriate birth control measures to ensure pregnancy will be excluded
* The patient has participated as a randomized patient in any investigational drug study within 30 days (starting from the final follow-up visit of that study) preceding the SV or plans to participate in another investigational drug study at any time during this study.
* The patient has a known hypersensitivity to any corticosteroid, salmeterol, or any of the excipients in the study drug (ie, lactose).
* The patient has a culture-documented or suspected bacterial or viral upper respiratory tract infection (URTI) or lower respiratory tract infection (LRTI), sinus, or middle ear that has not resolved at least 2 weeks before the SV.
* The patient has had an asthma exacerbation requiring systemic corticosteroids within 30 days before the SV, or has had any hospitalization for asthma within 2 months before the SV.
* The patient has used immunosuppressive medications within 4 weeks before the SV.
* The patient has untreated oral candidiasis at the SV. Patients with clinical visual evidence of oral candidiasis who agree to receive treatment and comply with appropriate medical monitoring may enter the study. Note: Azole antifungals are prohibited.
* The patient is an immediate relative of an employee of the investigational center.
* Patients who have donated whole blood 60 days before the first dose, or receive or donate plasma, white blood cells, or platelets within the 14 days before the first dose or study drug, and for 90 days after last dose of study drug.
* The patient has a disease/condition that in the medical judgment of the investigator would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.

  * Additional criteria apply, please contact the investigator for more information.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | 4 months
Area under the plasma drug concentration-time curve (AUCO-t) | 4 months

SECONDARY OUTCOMES:
Time to maximum observed plasma drug concentration (tmax) | 4 months

OTHER OUTCOMES:
Incidents of Participants with Adverse Events | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (3):
- United States (3):
  - Teva Investigational Site 13679, Huntington Beach, California
  - Teva Investigational Site 13678, Raleigh, North Carolina
  - Teva Investigational Site 13677, San Antonio, Texas